CLINICAL TRIAL: NCT06697886
Title: To Evaluate the Efficacy and Safety of Antiwei Granules in the Treatment of Common Cold (Wind-cold Syndrome) in a Multicenter, Randomized, Double-blind, Placebo-controlled Phase Ⅲ Clinical Trial
Brief Title: A Study of the Efficacy and Safety of Antiwei Granules in the Treatment of Common Cold
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-ATWKL-Ⅲ
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antaiwei granules (Experimental)
  Interventions: Drug: Antiwei Granules
- Antaiwei granules placebo (Placebo Comparator)
  Interventions: Drug: Antiwei Granules Placebo

INTERVENTIONS:
Drug: Antiwei Granules — During the 3-day treatment period, participants will receive 9 sacks of Antiwei granules. Oral administration, 1 sack (6g) per time, 3 times daily.
  Arms: Antaiwei granules
Drug: Antiwei Granules Placebo — During the 3-day treatment period, participants will receive 9 sacks of Antiwei granules. Oral administration, 1 sack (6g) per time, 3 times daily.
  Arms: Antaiwei granules placebo

SUMMARY:
To further evaluate the efficacy and safety of Antiwei granule in the treatment of common cold (wind-cold syndrome)

ELIGIBILITY:
Inclusion Criteria:

1. It met the diagnostic criteria of common cold in western medicine;
2. In accordance with the TCM syndrome differentiation standard of wind-cold syndrome;
3. Male and female patients aged 18 to 65 years;
4. The disease duration at enrollment was ≤48 h;
5. At enrollment, 37.3 ° C ≤axillary temperature < 38.5 ° C;
6. Informed consent was obtained voluntarily.

Exclusion Criteria:

1. Complicated with influenza, pneumonia, suppurative tonsillitis, acute tracheobronchitis, acute pharyngeal conjunctivitis, acute viral or herpetic pharyngitis, acute viral or herpetic laryngitis;
2. Patients who had been infected with 2019-ncov in the past and still had symptoms such as cough and fatigue for nearly 3 months after the antigen turned negative;
3. Primary ciliary dyskinesia syndrome, other acute onset nasal diseases (such as allergic rhinitis, chronic rhinitis, acute and chronic sinusitis, etc.), previous nasal surgery or radiotherapy of the nasopharynx with nasal mucosal dysfunction；
4. Patients with chronic respiratory diseases (such as chronic obstructive pulmonary disease, interstitial lung disease, etc.), asthma, and tuberculosis;
5. White blood cell count >12.0×10^9/L or <3.0×10^9/L , And/or neutrophil percentage >80%;
6. Aspartate aminotransferase and/or alanine aminotransferase ≥ 1.5 × ULN, or serum creatinine ≥ ULN, judged by the investigator to be clinically significant；
7. Combined with other serious primary diseases of the heart, brain, lung, liver, kidney or blood system, such as unstable control/serious complications of diabetes, viral hepatitis, hemophilia, or mental disorders;
8. Patients who had been treated with Chinese and western drugs for the relief of common cold and its symptoms after the onset of the current illness, including but not limited to antibiotics, antiviral, antihistamine, steroids, decongestants, antipyretic and analgesic, antitussive and expectorant drugs etc;
9. Those who were allergic to the known composition of the investigational drug or to emergency medication, or emergency drug contraindication population;
10. The participants (and their partners) had planned pregnancy or were unwilling to take appropriate contraceptive measures from enrollment to 1 month after the end of the trial, or were pregnant or lactating;
11. Suspected or true history of alcohol or drug abuse;
12. Participants who had participated in another clinical trial within 1 month before enrollment;
13. Persons deemed unsuitable for clinical trial by the investigator (e.g., athletes or persons not eligible for enrollment for other reasons).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
cure rate after 3 days of treatment | 3 days
  Disease recovery criteria: bad wind and cold, nasal congestion, runny nose, body pain, headache, sneezing, pharyngeal itching/sore throat symptoms were all relieved and body temperature to normal (axillary temperature < 37.3 ° C) and was maintained for at least 24 hours.
  Subjects were required to be treated before the first dose, D2-Cold-related symptoms since the last evaluation were evaluated in the morning and evening of D5 and in the morning of D6, respectively.

SECONDARY OUTCOMES:
Time to recovery | 3 days
  Disease recovery criteria: bad wind and cold, nasal congestion, runny nose, body pain, headache, sneezing, pharyngeal itching/sore throat symptoms were all relieved and body temperature to normal (axillary temperature < 37.3 ° C) and was maintained for at least 24 hours.
  Subjects were asked to evaluate their cold-related symptoms since the last evaluation before the first dose, in the morning and evening of D2-D5, and in the morning of D6. Visit 2 occurred on the morning of D6 after the assessment was completed.
  If the participant in visit 2 did not reach the recovery criteria according to the investigator's judgment, the diary card was reissued and the cold-related symptoms since the last evaluation were evaluated in the evening of D6, the morning and evening of D7, and the morning of D8
Remission rate after 3 days of treatment | 3 days
  Disease remission criteria: bad wind and cold, nasal congestion, runny nose, body pain, headache, sneezing, pharyngeal itching/sore throat were all asymptomatic or mild, and body temperature to normal (axillary temperature < 37.3 ° C) and was maintained for at least 24 hours.
  The ratio of subjects who achieved the remission standard after 3 days of medication was calculated, and whether the remission standard was reached was determined according to the morning and evening evaluation of D2-D5.
Single symptom disappearance rate after 3 days of medication | 3+1 days
  Single symptoms included bad wind and cold, nasal congestion, runny nose, body pain, headache, sneezing, pharyngeal itching/sore throat .
  Single symptom disappearance was defined as the disappearance of each single symptom (axillary temperature < 37.3℃) and maintained for at least 24 hours.
Efficacy of TCM syndrome after 3 days of medication | 3 days
  After 3 days of treatment, the proportion of subjects who were cured/better/effective in each group was calculated.Clinical recovery: clinical symptoms and signs basically disappeared or completely disappeared, and the syndrome score decreased by ≥95% compared with the baseline. Marked effect: the clinical symptoms and signs were significantly improved, and the syndrome score was reduced by ≥70% compared with the baseline. Effective: the clinical symptoms and signs were improved, and the syndrome score decreased by ≥30% compared with the baseline; No effect: the clinical symptoms and signs did not change, or even had a trend of aggravation, and the syndrome score decreased less than 30% compared with the baseline.
Changes in single symptom level after 3 days of medication | 3 days
  The change of each symptom score from baseline to 3 days after treatment was calculated.
  Single symptom: bad wind and cold, nasal congestion, runny nose, body pain, headache, fever, sneezing, pharyngeal itching/sore throat, cough, fatigue.
Incidence of complications | 3 days
  The proportion of subjects with complications (including acute sinusitis, otitis media, tracheobronchitis, pneumonia, etc.) during the period from the first administration of the trial drug to the completion of the trial was calculated.
Proportion of subjects using emergency medication | 3 days
  If the subject's body temperature (axillary temperature) exceeds 39 ° C during the trial, If the body temperature reaches 38.5℃ or above for 4 hours, or if the patient cannot tolerate it, temporary acetaminophen tablets can be taken according to the doctor's advice.
The cure rate of cough and all cold symptoms after 3 days of treatment | 3 days
  Cough and all cold symptoms recovery criteria: cough, bad wind and cold, nasal congestion, runny nose, body pain, headache, sneezing, pharyngeal itching/sore throat symptoms were all relieved and body temperature to normal (axillary temperature < 37.3 ° C) and was maintained for at least 24 hours.

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - Beijing Hospital of Traditional Chinese Medicine, Capital Medical University, Beijing
  - changsha Hospital Affiliated to Hunan University, Changsha
  - Chengdu Pidu District Hospital of TCM, Chengdu
  - Heilongiang Provincial Traditional Chinese Medicine Hospital, Haerbin
  - The Second Affiliated Hospital of Heilongjiang University of Chinese Medicine, Haerbin
  - Huizhou Third People's Hospital, Huizhou
  - Kaifeng Hospital of Traditional Chinese Medicine, Kaifeng
  - Luoyang Third People's Hospital, Luoyang
  - The Affiliated Traditional Chinese Medicine Hospital, Southwest Medical University, Luzhou
  - The Affiliated Hospital of Jiangxi Uniwersity of TCM, Nanchang
  - Panjin Liaoyou Baoshihua Hospital, Panjin
  - Quzhou People's Hospital, Quzhou
  - Sanmenxia Central Hospital, Sanmenxia
  - Longhua Hospital, Shanghai University of Traditional Chinese Medicine,, Shanghai
  - Shangqiu First People's Hospital, Shangqiu
  - The Second Affiliated Hospital of Liaoning University of Traditional Chinese Medcine, Shenyang
  - Hebei Provincial Hospital of Traditional Chinese Medicine, Shijiazhuang
  - The Second Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin
  - Tonghua Central Hospital, Tongzhou
  - The Second Affiliated Hospital of Shaanxi University of Chinese Medicine, Xi'an
  - Xidian Group Hospital, Xi'an
  - The Second Affiliated Hospital of Xingtai Higher Medical College, Xingtai
  - Yangquan Coal Industry(Group) General Hospital, Yangquan
  - Henan Provincial People's Hospital, Zhengzhou